CLINICAL TRIAL: NCT01334580
Title: Comparison of Cognitive-Behavioral Therapy and Methadone Drug Counseling for Methadone-Maintained Patients With Co-occurring Chronic Pain and Opioid Dependence
Brief Title: Cognitive-Behavioral Therapy for Pain and Opioid Dependence in Methadone Maintenance Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 0703002496_B; K23DA024050-03 (NIH)
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Chronic Pain; Opiate Dependence
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methadone Drug Counseling (Active Comparator): Methadone Drug Counseling is provided by skilled drug counselors over a 12 week period and focuses on cessation of illicit drugs
  Interventions: Behavioral: Methadone Drug Counseling
- Cognitive-Behavioral Therapy for Pain and Opioid Dependence (Experimental): CBT is provided by skilled psychologists in weekly sessions for 12 weeks and focuses on reducing illicit drug use and increasing pain management.
  Interventions: Behavioral: Cognitive-Behavioral Therapy for Pain and Opioid Dependence

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy for Pain and Opioid Dependence — CBT is provided by skilled psychologists in weekly sessions for 12 weeks and focuses on reducing illicit drug use and increasing pain management.
  Arms: Cognitive-Behavioral Therapy for Pain and Opioid Dependence
Behavioral: Methadone Drug Counseling — Methadone Drug Counseling (MDC)is provided by skilled drug counselors over a 12-week period. The primary goal of MDC is cessation of illicit drugs.
  Arms: Methadone Drug Counseling

SUMMARY:
This study involves the comparison of two treatment approaches for patients with chronic pain who are entering methadone maintenance treatment (MMT) for opioid addiction: (a) an integrated counseling that addresses both chronic pain and opioid dependence(POD)and (b) a counseling intervention that addresses opioid dependence only.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* prescription opioid or heroin addiction
* moderate to severe chronic pain
* enrolled in methadone maintenance at the APT Foundation for opioid addiction
* understand English

Exclusion Criteria:

* current suicide or homicide risk
* life-threatening or unstable medical problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Pain reduction | 16 weeks
Reduce illicit opioid use | 16 weeks

SECONDARY OUTCOMES:
Finalization of treatment manuals | 16 weeks
Development and modification of therapy training and process rating measures | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Declan Barry, PhD, Principal Investigator — Yale University
Locations (1):
- Methadone Research Unit, New Haven, Connecticut, United States